CLINICAL TRIAL: NCT07003815
Title: A Single-Arm, Exploratory Clinical Study of Envafolimab Combined With Gemcitabine, Cisplatin, and Simvastatin for the Treatment of Locally Advanced or Metastatic BTC Patients
Brief Title: Envafolimab With Chemotherapy and Simvastatin in Advanced Biliary Tract Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Wan-Guang Zhang, Chief Physician, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB202401114
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Biliary Tract Cancer; Advanced Cancer
Keywords: Biliary Tract Cancer; Envafolimab; Simvastatin; Immunotherapy; Chemotherapy
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — envafolimab; Gemcitabine; Cisplatin; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Envafolimab + Gemcitabine/Cisplatin + Simvastatin Combination Therapy (Experimental): Intervention(s):
  All enrolled participants will receive the following combination therapy:
  Envafolimab (300 mg, intravenous infusion, Day 1 of each 21-day cycle) - a PD-L1 inhibitor immunotherapy.
  Gemcitabine (1,000 mg/m², IV, Days 1 and 8 of each cycle) + Cisplatin (25 mg/m², IV, Days 1 and 8 of each cycle) - standard chemotherapy regimen.
  Simvastatin (40 mg, oral daily) - repurposed as a potential synergistic agent.
  Treatment Schedule:
  Initial Phase (Cycles 1-8):
  21-day cycles for up to 8 cycles (≈6 months). Drugs administered as above.
  Maintenance Phase (Post-Cycle 8):
  Continue Envafolimab (300 mg, IV, every 28 days) + Simvastatin (40 mg, oral daily) until disease progression or unacceptable toxicity.
  Interventions: Drug: Envafolimab + Gemcitabine + Cisplatin + Simvastatin

INTERVENTIONS:
Drug: Envafolimab + Gemcitabine + Cisplatin + Simvastatin — Envafolimab (generic name):
  Dose: 300 mg, intravenous (IV) infusion. Schedule: Day 1 of each 21-day cycle (induction phase); every 28 days (maintenance phase).
  Role: PD-L1 inhibitor immunotherapy.
  Gemcitabine (generic name):
  Dose: 1,000 mg/m², IV infusion. Schedule: Days 1 and 8 of each 21-day cycle (induction phase only).
  Cisplatin (generic name):
  Dose: 25 mg/m², IV infusion. Schedule: Days 1 and 8 of each 21-day cycle (induction phase only).
  Simvastatin (generic name):
  Dose: 40 mg, oral tablet. Schedule: Daily (continuously through induction and maintenance phases). Investigational Role: Potential immunomodulator and chemosensitizer in biliary tract cancer.
  Treatment Phases:
  Induction Phase (Cycles 1-8, 21-day cycles): All four drugs administered. Maintenance Phase (Post-Cycle 8): Envafolimab + Simvastatin only (28-day cycles).

SUMMARY:
Brief Summary

The goal of this clinical trial is to test whether the combination of Envafolimab (an immunotherapy drug), chemotherapy (gemcitabine + cisplatin), and simvastatin can help treat advanced biliary tract cancer (BTC) that cannot be removed by surgery or has spread. The study will also evaluate the safety of this treatment combination.

Key Questions Does the combination treatment help shrink tumors or slow cancer growth better than standard options? What side effects do participants experience with this treatment?

What Will Participants Do? Receive Envafolimab (IV infusion) + gemcitabine/cisplatin (chemotherapy) + simvastatin (oral pill) every 3 weeks for up to 8 cycles (~6 months).

After 8 cycles, continue with Envafolimab + simvastatin alone every 4 weeks until cancer worsens or side effects become too severe.

Undergo regular scans, blood tests, and clinic visits to monitor tumor response and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age : ≥18 years old.
* Diagnosis : Histologically confirmed unresectable, locally advanced, or metastatic biliary tract adenocarcinoma (including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, and gallbladder cancer).
* Prior Treatment :Treatment-naïve for unresectable/metastatic disease at initial diagnosis, OR Disease recurrence ≥6 months after curative surgery or adjuvant therapy.
* Performance Status : ECOG PS 0 or 1.
* Measurable Disease : At least one radiologically measurable lesion per RECIST 1.1 (tumor lesion ≥10 mm on CT scan, lymph node ≥15 mm in short axis).
* Organ Function : No severe functional impairment of heart, lung, brain, or other vital organs.

Exclusion Criteria:

* Disease Type : Ampulla of Vater cancer.
* Autoimmune Disease : Active or previously documented autoimmune/inflammatory disorders.
* Allergy : Hypersensitivity to any study drug (Envafolimab, gemcitabine, cisplatin, or simvastatin).
* Liver Function : Decompensated liver dysfunction.
* Psychiatric History : Severe psychiatric disorders.
* Recent Trials : Participation in other drug/device trials within 4 weeks prior to enrollment.
* Compliance : Inability to adhere to protocol requirements or follow-up schedule.
* Investigator's Discretion : Any other condition deemed unsuitable for participation by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) at 24 Weeks | From treatment initiation until 24 weeks (or disease progression, if earlier).
  Proportion of participants achieving complete response (CR) or partial response (PR) per RECIST 1.1 criteria, assessed by CT/MRI scans after 24 weeks of treatment. CR: disappearance of all target lesions; PR: ≥30% decrease in target lesion diameters.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 2 years.
  Time from treatment start to disease progression (per RECIST 1.1) or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to 2 years.
  Time from treatment start to death from any cause.
Disease Control Rate (DCR) | Up to 2 years.
  Proportion of participants with CR, PR, or stable disease (SD) lasting ≥12 weeks.
Duration of Response (DOR) | Up to 2 years.
  Time from first documented response (CR/PR) to disease progression or death.
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From first dose until 30 days after last dose.
  Frequency and severity of adverse events graded by CTCAE v5.0.